CLINICAL TRIAL: NCT03651505
Title: X-linked Hypophosphatemia Disease Monitoring Program (XLH-DMP)
Brief Title: X-linked Hypophosphatemia Disease Monitoring Program
Status: Active, not recruiting | Type: Observational
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: UX023-CL401
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: X-linked Hypophosphatemia; Hypophosphatemic Rickets
Keywords: X-linked Hypophosphatemia; Fibroblast growth factor 23 (FGF23); KRN23; XLH; Hypophosphatemia; Familial Hypophosphatemic Rickets; FGF23; Crysvita
MeSH Terms: conditions — Familial Hypophosphatemic Rickets; Rickets, Hypophosphatemic; Hypophosphatemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prior Burosumab Clinical Trial Participants: Patients who participated in burosumab clinical trials and continue to receive burosumab via prescription from their physician.
  Interventions: Other: No intervention
- Not from Prior Burosumab Clinical Trial: Patients may take other treatments for XLH and may start burosumab treatment at any time as prescribed by a physician.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Access to any treatment is through authorized commercial use and not as a part of this DMP

SUMMARY:
The objectives of this observational study are to characterize XLH disease presentation and progression and to assess long-term effectiveness and safety of burosumab.

DETAILED DESCRIPTION:
The XLH-DMP is a global, prospective, multicenter, longitudinal, long-term outcomes program for subjects on or off any treatment designed to characterize XLH disease presentation and progression, assess long-term safety and effectiveness of burosumab, as well as prospectively investigate longitudinal change over time across biomarker(s), clinical assessments, and patient/caregiver-reported outcome measures in a representative population. The XLH-DMP will collect demographic, biochemical, physiologic, disease severity, and progression data in patients taking burosumab and those not taking burosumab. In this DMP, patients will only have access to burosumab through authorized prescribed use. The Sponsor will not provide any treatments as part of the DMP.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent or, in the case of patients under the age of 18 years (or 16 years, depending on the region), provide assent (if required) and informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Clinical diagnosis of XLH based on family history, OR confirmed PHEX mutation, OR biochemical profile consistent with XLH.
* Willing and able to comply with the study visit schedule and study procedures.

Exclusion Criteria:

* Concurrent enrollment in an Ultragenyx-sponsored clinical trial is NOT permitted.
* Serious medical or psychiatric comorbidity.
* Less than one year of life expectancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 800 eligible adult and pediatric patients with XLH will be enrolled globally, with a minimum of 200 pediatric patients. Patients can enter the XLH-DMP regardless of how their XLH is being treated. Patients on Crysvita (burosumab) via prescription may begin taking Crysvita, per standard of care before or after enrolling in the XLH DMP.
Sampling Method: Non-Probability Sample
Enrollment: 782 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Long-Term Safety of Burosumab | 10 years
  To assess the long-term safety of burosumab treatment in adult and pediatric patients with XLH, including overall renal health, the presence and/or progression of nephrocalcinosis and spinal stenosis, and pregnancy outcomes.
Long-Term Effectiveness of Burosumab | 10 years
  To evaluate the long-term effectiveness of burosumab treatment on key manifestations of XLH, including skeletal health, stiffness, mobility and physical functioning.
Clinical Course of XLH Disease | 10 years
  To illustrate the clinical, radiological, biochemical manifestations and progression of XLH over time in both untreated and treated patients with XLH.

CONTACTS AND LOCATIONS:
Overall Officials: Ultragenyx Medical Director, Study Director — Ultragenyx Pharmaceuticals Inc.
Locations (38):
- United States (24):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University - Department of Medicine, Nashville, Tennessee
  - Vanderbilt University - Department of Pediatrics, Nashville, Tennessee
  - Houston Methodist Research Institute, Houston, Texas
  - University of Texas, Health Science Center, Houston, Texas
  - University of Virgina School of Medicine, Charlottesville, Virginia
  - Children's Hospital of The King's Daughter, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - American Family Children's Hospital, Madison, Wisconsin
- Argentina (3):
  - Hospital General de Niños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D.
  - Hospital de Niños Dr. Ricardo Gutierrez, Buenos Aires
  - Hospital Privado Universitario de Córdoba, Córdoba
- Brazil (4):
  - Hospital Universitário Alcides Carneiro (HUAC), São José, Campina Grande - PB
  - Instituto de Medicina Avancada (IMA Brasil), São Paulo, São Paulo
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
- Canada (4):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Bone Research and Education Centre, Oakville, Ontario
  - Shiner's Hospital for Children - Canada, Montreal, Quebec
  - Children's Hospital Eastern Ontario Research Institute, Ottawa
- Pontificia Universidad Católica de Chile, Santiago, Santiago Metropolitan, Chile
- Colombia (2):
  - Hospital Universitario de San Vicente Fundación, Medellín, Antioquia
  - Hospital Infantil Universitario de San José, Bogotá, Cundinamarca

REFERENCES:
- [Derived] Carpenter TO, Fukumoto S, Haffner D, Imel EA, Ozono K, Ishii H, Li Z, Sandilands K, Joos-Vandewalle P, Lee C, Kanematsu M, McCullough KP, Brandi ML. Advancing Patient Evidence in XLH (APEX): Baseline analysis of a global data unification program. Bone. 2025 Dec;201:117649. doi: 10.1016/j.bone.2025.117649. Epub 2025 Sep 15. PMID 40962182
- See also: Ultragenyx Transparency Commitment — http://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/